CLINICAL TRIAL: NCT01205425
Title: Role of Computed Tomography Coronary Angiography in Optimalization of Percutaneous Coronary Interventions With Stent Implantation.
Brief Title: Computed Tomography Coronary Angiography Before Stent Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Collaborators: Ministerstwo Nauki i Szkolnictwa Wyższego, Warszawa, Polska (Unknown)
Responsible Party: Jerzy Pregowski, Institute of Cardiology, 04-628 Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: N N403 295736
Record Dates: First submitted 2010-06-25; First posted 2010-09-20 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Stable Coronary Artery Disease
Keywords: Computed coronary angiography; Stent implantation; IVUS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- CT (Experimental): Procedure of stent implantation will be planed on the basis of both angiography and computed tomography results.
  Interventions: Procedure: CT guided PCI
- Angio (Active Comparator): Procedure of stent implantation will be planned only on the basis of diagnostic coronary angiography.
  Interventions: Other: PCI on the basis of coronary angiography

INTERVENTIONS:
Other: PCI on the basis of coronary angiography — Interventional cardiologist will be blinded to the images obtained by CT. The PCI procedure will be planned and performed solely on the basis of invasive coronary angiography
  Arms: Angio
Procedure: CT guided PCI — The results of the CT scan will be analysed by the interventional cardiologist that is to perform angiography and PCI. Based on this analysis preliminary procedural strategy is planned (stent diameters, decision on direct stenting vs. predilatation, decision on postdilation)
  Arms: CT

SUMMARY:
The purpose of the study is to determine whether results of the computed tomography coronary angiography may be helpful in planning and performing percutaneous angioplasty in patients with stable angina pectoris.

DETAILED DESCRIPTION:
Currently most percutaneous coronary interventions (PCI) are planned and performed on the basis of invasive coronary angiography which provides the information that is confined to the vessel lumen. This limitation may be partially responsible for the unfavorable long term outcome and complications that occur in some patients. Additional information on the disease burden in angiographically normal coronary segments adjacent to the lesion site could impact the treatment strategy and clinical results. Imaging modalities that allow not only lumen but also vessel wall assessment include both invasive (e.g. intravascular ultrasounds - IVUS) and non-invasive (e.g. multislice computed tomography - MSCT) methods. IVUS guidance of the coronary interventions is expensive and given its invasiveness is related to the additional risk. The number of patients who are referred for coronary angiography with significant stenosis diagnosed with MSCT is rapidly increasing. Most interventional cardiologists are not familiar with coronary vessel images produced by MSCT. The aim of our study is to assess if the analyses of MSCT images before the PCI may impact the treatment strategy and immediate results. The study will enroll subjects with significant coronary stenosis diagnosed with MSCT who are referred to the catheterisation laboratory for invasive angiography and PCI. The study participants will be randomized into two groups:

Group 1 - the results of MSCT are analysed by the interventional cardiologist that is to perform angiography and PCI. Based on this analysis preliminary procedural strategy is planned (stent diameters, decision on direct stenting vs. predilatation, decision on postdilation) Group 2 - interventional cardiologist is blinded to the images obtained by MSCT. The PCI procedure is performed solely on the basis of invasive coronary angiography In both study groups IVUS will be performed before and after stent implantation. The operator will be blinded to the results of pre-PCI IVUS. The second IVUS will be performed when angiographic results are optimal in the opinion of the operator. The results of the second IVUS examination will be the efficacy measure of the two compared treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Stable coronary artery disease
* Planned stent implantation into single lesion in native coronary artery
* Planned stent diameter: 2.5-4.0 mm

Exclusion Criteria:

* Women younger than 50 years
* Lesion location in left main coronary artery
* Atrial fibrilation or other significant arrythmia
* Severe chronic obturatory pulmonary disease
* Hyperthyroidism
* Known allergy to contrast media
* Glomerular filtration rate < 30
* Treatment of bifurcation lesion
* Stent implantation for in-stent restenosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Minimal in stent lumen area as assessed by IVUS | Up to 10 minutes after stent implantation
Adequacy of lesion coverage defined as minimal lumen area in reference segments adjacent to stent shoulder. | Up to 10 minutes after stent implantation

SECONDARY OUTCOMES:
Mean stent lumen area | Up to 10 minutes after stent implantation
Mean lumen area and plaque and media area in 10mm segments adjucent to stent edges. | Up to 10 minutes after stent implantation
Qualitative and quantitative assessment of potential complications (tissue prolaps, plaque shift, stent edge dissection and stent malapossition) | Up to 10 minutes after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Jerzy Pregowski, MD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- See also: Web page of Institute of Cardiology, Warsaw — http://www.ikard.pl